CLINICAL TRIAL: NCT01008800
Title: Parent-mediated vs Center-based Intervention for Toddlers With ASD: An RCT
Brief Title: A Randomized Clinical Trial for Toddlers With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Landa, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R40 MC 15594-01; NA_00030329 (Other: Johns Hopkins Medicine IRB #)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; language; social; toddlers
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Center-Based classroom intervention (Experimental): Four days a week for 2.5 hours a day the child will participate in a classroom with peers in an attempt to increase social communication, language abilities, and other skills. Parents will also receive education sessions 1-3 times per month for 1-2 hours each. Treatment will last for 6 months.
  Interventions: Behavioral: Social Communication
- Parent Training (Active Comparator): Parents are taught strategies on how to interact with their children to increase their skills. Parent training sessions are given 2 times a month at our center and once a month at home for 60-90 minutes each. Treatment will last for 6 months.
  Interventions: Behavioral: Social communication

INTERVENTIONS:
Behavioral: Social Communication — The Center-Based classroom intervention focuses on providing children with an invigorating, motivating learning environment in which emerging skills and knowledge are skillfully brought to a higher level of maturity, integrated with existing abilities, and used functionally. Providing an enriched environment with toys, structured learning, and opportunities for ongoing engagement week may offer the children experiences that they would not otherwise have (Ramey & Ramey, 1998). Parent training sessions will focus on strategies aimed at improving child social engagement and communication and on topics related to autism characteristics, learning styles, interventions, and resources.
  Arms: Center-Based classroom intervention
Behavioral: Social communication — Parent training sessions will focus on teaching parents strategies for enhancing their child's social engagement and communication. Since parents will be using these strategies across all activities throughout the day, there is an increased likelihood of generalization. For parents of minority and underserved children, this may be the first exposure to responsive interaction strategies (Rudy & Grusec, 2001).
  Arms: Parent Training

SUMMARY:
This research is being done to test the effectiveness of two treatments aimed at increasing language and social skills in children with autism spectrum disorder. If children show improvement in these treatments, we hope that the availability of public services for minority and low income families will be increased. Minority and low income families with children between 22 and 33 months of age with Autism Spectrum Disorders may join.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 22 to 33 months old
* Children must meet criteria for ASD or autism on the ADOS plus receive a clinical judgment of PDD-NOS or autism by the study team
* Children must have an age equivalent of 8 months or greater for non-verbal ability based on the Mullen Visual Reception and Fine Motor scales
* Parents must agree to participate in the study and commit to having their child participate in the intervention to which they are randomized for 6 months
* The parent (or other primary caregiver, such as grandparent) in the Parent-Mediated condition must agree to attend the training sessions three times per month
* Parents must be between the ages of 16 and 50 years old
* Families who qualify for medical assistance and/or have racial/ethnic minority backgrounds will be prioritized for recruitment and participation in this study. On the TSI, we will ask participants if they qualify for medical assistance or if they are of a racial minority or have a first degree relative of a racial minority. Families who do not fit these criteria will be notified that they may be eligible to participate if additional space is available.
* It is not required that English be their primary language, but they must be fluent in English (or if the child is nonverbal he/she must hear English most of the time at home)

Exclusion Criteria:

* Head injury prior to enrollment in the study
* Major hearing or visual impairment after correction
* Non-febrile seizures
* PKU (Phenylketonuria)
* Congenital Rubella (German measles)
* Neurofibromatosis
* Tuberous Sclerosis
* Fragile X
* A fall resulting in a loss of consciousness or other severe head injury
* Velo-Cardio Facial Syndrome
* Any other known genetic syndrome
* No foster children may participate
* The child must not be adopted

Ages: 22 Months to 33 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Communication and Symbolic Behavior Scales | immediately after treatment ends and 6 months after treatment ends

SECONDARY OUTCOMES:
Mullen Scales of Early Learning | immediately after treatment ends and 6 months after treatment ends

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Sofronoff K, Farbotko M. The effectiveness of parent management training to increase self-efficacy in parents of children with Asperger syndrome. Autism. 2002 Sep;6(3):271-86. doi: 10.1177/1362361302006003005. PMID 12212918
- [Background] Tannock R, Girolametto L, Siegel LS. Language intervention with children who have developmental delays: effects of an interactive approach. Am J Ment Retard. 1992 Sep;97(2):145-60. PMID 1384566
- [Background] McGee, G. G., Morrier, M. J., & Daly,T. (1999).An incidental teaching approach to early intervention for toddlers with autism. Journal of the Association for Persons with Severe Handicaps, 24, 133-146.
- [Background] Rutter M. Diagnosis and definition of childhood autism. J Autism Child Schizophr. 1978 Jun;8(2):139-61. doi: 10.1007/BF01537863. No abstract available. PMID 670129
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638